CLINICAL TRIAL: NCT07101432
Title: Phase I Study of Preconditioning Radiation Therapy With IL-15 Transduced TGFBR2 KO CAR.TROP2-engineered Cord Blood-derived NK Cells in Patients With Advanced Head and Neck Cancer (RADIANCE-NK)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0561; NCI-2025-05464 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 ESC Safety Lead-in - TROP2 CAR/IL-15 TGFBR2 KO NK Cells (Experimental): Participants will receive treatment on an outpatient basis
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 ESC/EXP - TROP2 CAR/IL-15 TGFBR2 KO NK Cells + RT (Experimental): Participants will receive treatment on an outpatient basis
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine — Given by infusion
Drug: Cyclophosphamide — Given by infusion

SUMMARY:
To find the recommended dose of an investigational therapy called chimeric antigen receptor (CAR).TROP2/interleukin (IL)15-transduced TGFBR2 KO cord blood (CB)-derived natural killer (NK) cells (TROP2 CAR/IL-15 TGFBR2 KO NK cells) that can be given with and without preconditioning radiation therapy in patients with advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety, tolerability, and recommended Phase 2 dose (RP2D) of chimeric antigen receptor (CAR).TROP2/interleukin (IL)15-transduced TGFBR2 KO cord blood (CB)-derived natural killer (NK) cells (TROP2 CAR/IL-15 TGFBR2 KO NK cells) combined with and without preconditioning RT in patients with advanced head and neck squamous cell carcinoma.

Secondary Objectives:

1. To determine the antitumor activity of TROP2 CAR/IL-15 TGFBR2 KO NK cells, including those with pre-CAR-NK bridging SBRT in patients eligible to receive this. Although the clinical benefit of TG TROP2 CAR/IL-15 TGFBR2 KO NK cells has not yet been established (and is currently being investigated in other solid tumors in other clinical trials we have rendered), the intent of offering this treatment is to provide a possible therapeutic benefit and thus, the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability. Efficacy will be determined in each cohort, and for this, we will have a pre-planned subset analysis of patients with metastatic disease where one site is not irradiated.
2. To quantify the persistence of infused allogeneic donor CAR-transduced CB-derived NK cells in the peripheral blood of the recipient.
3. To conduct comprehensive immune modulation studies by evaluating tissue and bloodbased biomarkers associated with response and resistance to TROP2 CAR/IL-15 TGFBR2 KO NK cell infusion.
4. To obtain preliminary data on quality of life and patient experience.
5. To evaluate longitudinal changes in circulating tumor DNA (ctDNA).

Exploratory Objectives:

1. In patients who do not receive SBRT due to ineligibility, they are still eligible to receive CAR-NK cell therapy. This inadvertent biologic randomization may enable cross-sectional comparison of outcomes and correlatives among the patients who receive RT vs. not.
2. To quantify the progression-free survival, overall survival, and the duration of responses of TGFBR2 KO CAR.TROP2/IL15-transduced CB-derived NK cells combined with preconditioning RT in patients with advanced head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically confirmed head and neck cancer, either HPV+ or HPV-, that is locally advanced AND unresectable OR metastatic (≤5 sites of disease), which has relapsed or progressed following local standard treatments that are known to prolong survival, or for which no standard treatment is available or are no longer effective, or refused such therapy.

Patient tumors must demonstrate TROP2 expression of 2+ or 3+ as determined by IHC at the MDACC CAP and CLIA accredited Clinical Laboratories.

* 2 weeks from the last cytotoxic chemotherapy at the time of lymphodepleting chemotherapy; ≥3 days from last TKI or other targeted therapies at the time of lymphodepleting chemotherapy; ≥3 months from any cell therapy for any malignancy at the time of lymphodepleting chemotherapy; prior radiation therapy is allowed at the time of consent.

RT allowed to ≥1 disease sites prior to the lymphodepleting chemotherapy. If there are additional measurable non-irradiated disease sites, this may be evaluated for response as well. If multiple lesions are irradiated, we advise that a single lesion will be treated to a higher dose and other lesions considered for lower doses, and that one site always remain unirradiated if a patient has ≥2 sites of disease.

Age ≥18 years. Because no dosing or adverse event data are currently available on the use of TROP2 CAR/IL-15 TGFBR2 KO NK cells in combination with radiation therapy in patients <18 years of age, children are excluded from this study.

Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Life expectancy ≥3 months per PI or treating physician's discretion.

A female patient is eligible to participate if at least one of the following conditions applies:

a. Not a woman of childbearing potential (WOCBP). OR

A WOCBP who agrees to follow the contraceptive guidelines in Appendix 5 during the study treatment period and for 6 months post-TROP2 CAR/IL-15 TGFBR2 KO NK cell infusion.

WOCBP must have a negative urine pregnancy test within 72 hours prior to the start of lymphodepleting chemotherapy. If a WOCBP has a urine pregnancy test that cannot be confirmed as negative, a serum (beta-human chorionic gonadotropin [B-hCG]) pregnancy test will be required.

The effects of TROP2 CAR/IL-15 TGFBR2 KO NK cells on the developing human fetus are unknown. Radiation therapy is absolutely contraindicated in pregnant women. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

A female patient who becomes pregnant, or suspects pregnancy while she or her partner is participating in this study, must immediately notify her doctor. Female patients who become pregnant will be taken off study.

Male patients treated or enrolled on this protocol must agree to follow the contraceptive guidelines in Appendix 5 prior to study entry and for the duration of study participation and for 6 months post-TROP2 CAR/IL-15 TGFBR2 KO NK cell infusion. Male patients who father a child or suspect that they have fathered a child must immediately notify their doctor.

Patients must have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Patients must have adequate organ function as defined below within 10 days prior to the start of lymphodepleting chemotherapy:

Table 1. Adequate Organ Function Laboratory Values

Systemic Function Test Laboratory Value Hematologic ANC ≥ 1500/µL Platelets ≥ 100,000/µL Hemoglobin ≥9.0 g/dLa Renal Creatinine ≤ 1.5 x ULNb OR CrCl by Cockcroft-Gault ≥30 mL/min for patients with creatinine formula > 1.5 x ULNb Hepatic Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 x ULN AST and ALT ≤2.5 x ULN (≤5 x ULN for patints with liver metastases) Coagulation PT/INR ≤1.5 x ULN unless patien is receiving anticoagulant aPTT therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT=alanine aminotransferase; ANC=absolute neutrophil count; aPTT=activated partial thromboplastin time; AST=aspartate aminotransferase; CrCl=creatinine clearance; INR=international normalized ratio; PT=prothrombin time; ULN=upper limit of normal.

1. Criteria must be met without erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks of the screening test. Patients may be on a stable dose of erythropoietin (≥ approximately 3 months).
2. Serum creatinine and CrCl should be interpreted and calculated per institutional standard.

   Left ventricular ejection fraction >50%.

   Adequate respiratory reserve defined as dyspnea Grade 0 or 1 and saturated oxygen >92% in room air. See Table 2 for a grading scale of dyspnea per the CTCAE v5.0.

   Table 2. Dyspnea grading scale.

   Grade 0 - No shortness of breath Grade 1 - Shortness of breath with moderate exertion Grade 2 - Shortness of breath with minimal exertion; limiting instrumental ADL Grade 3 - Shortness of breath at rest; limiting self-care ADL Grade 4 - Life threatening consequences; urgent intervention indicated Grade 5 - Death

   Prior treatment with TROP2-targeted therapy will be allowed.

   Willing to undergo mandatory blood collections and biopsies as required by the study.

   Willing to sign consent for long-term follow-up on protocol PA17-0483.

   Willing to stay within a 2-hour drive (approximately 100-mile radius) of the study site during the first 4 weeks after the TROP2 CAR/IL-15 TGFBR2 KO NK cell infusion.

   Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

   Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

   Ability to understand and the willingness to sign a written informed consent document.

   Exclusion Criteria:
   1. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 6 months post TROP2 CAR/IL-15 TGFBR2 KO NK cell infusion.
   2. Has received systemic anticancer therapy within 2 weeks or 5 half-lives, whichever is shorter, prior to the start of lymphodepleting chemotherapy. For patients treated with monoclonal antibodies, at least 3 weeks must have elapsed prior to the start of lymphodepleting chemotherapy. Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
   3. Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI)/co-PIs. If a patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to the start of lymphodepleting chemotherapy.
   4. If patients receive RT within 2 weeks of the start of lymphodepleting chemotherapy, they must not require corticosteroids, and not have had radiation pneumonitis.
   5. Has received a live vaccine within 6 weeks prior to TROP2 CAR/IL-15 TGFBR2 KO NK infusion and for at least 24 months post infusion. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
   6. Prior CAR T or NK cell or other genetically modified T or NK cell therapy.
   7. Has diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent).
   8. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to patients who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
   9. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate if they completed radiation therapy, are clinically stable, and without requirement of steroid treatment for at least 2 weeks prior to study enrollment.
   10. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
   11. History of interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD. 12. Active infection requiring systemic therapy.

   13. Known human immunodeficiency virus (HIV) infection.

   14. Known active or chronic hepatitis B or hepatitis C virus infection.

   15. Known history of active tuberculosis (Mycobacterium tuberculosis).

   16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.

   17. Patients with psychiatric illness/social situations that would limit compliance with study requirements.

   18. Has had an allogenic tissue/solid organ transplant.

   19. Clinically significant cardiovascular disease within 12 months prior to the start of lymphodepleting chemotherapy, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebrovascular event, or cardiac arrhythmia associated with hemodynamic instability. NOTE: medically controlled arrhythmia would be permitted.

   20. Prolongation of corrected QT interval using Fridericia's formula to >480 milliseconds.

   21. Patients with bleeding or thrombotic disorders or at risk for severe hemorrhage. Patients with known deep vein thrombosis/pulmonary embolism who are on appropriate anti-coagulation treatment are eligible.

   22. Patients with history of ≥Grade 3 stomatitis or mucositis with prior therapy.

   23. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide and fludarabine or other agents used in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gohar Manzar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org